CLINICAL TRIAL: NCT00265473
Title: hOKT3γ1 (Ala-Ala), Sirolimus and Low Dose Tacrolimus Therapy in Type 1 Diabetic Islet Allograft Recipients
Brief Title: MGA031, Sirolimus and Tacrolimus in Islet Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0407M62505
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Results first posted 2011-09-21 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Allogeneic Islets of Langerhans (Experimental): Islet infusion
  Interventions: Biological: Allogeneic Islets of Langerhans

INTERVENTIONS:
Biological: Allogeneic Islets of Langerhans — Intraportal infusion of islets of Langerhans

SUMMARY:
This clinical trial is designed to extend the observations made in our pilot clinical trial (IND 8971, Study #1) on the safety and efficacy of immunotherapy with the anti-CD3 monoclonal antibody hOKT3γ1 (Ala-Ala), (currently called MGA031) combined with sirolimus and tacrolimus in preventing rejection and autoimmune destruction of deceased donor pancreatic islet transplants in type 1 diabetic recipients.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus continues to be a therapeutic challenge. Previous studies have shown that failure to prevent hypoglycemia and hyperglycemia results in acute and chronic complications, leading to poor quality of life, premature death, and considerable health care costs in 30% to 50% of diabetic patients. Therefore, establishing safe and effective ways to achieve and maintain normoglycemia would have substantial implications for the well-being of individuals with diabetes. Intensive insulin therapy has been shown to reduce the risk of chronic complications in patients who achieve near-normalization of glycemia. However, such therapy is labor-intensive, difficult to implement for many patients, and limited by the accompanying increased frequency of severe hypoglycemia. Currently, the only way to restore and sustain normoglycemia without the associated risk of hypoglycemia is by replacing the patient's islets of Langerhans, either by transplanting a vascularized pancreas or, much less invasively, by infusing isolated islets.

Strategies that selectively inactivate autoreactive T cells and prevent allorejection of transplanted islets in the absence of diabetogenic side effects need to be developed for islet transplants to survive in autoimmune diabetic recipients. The current clinical study will extend the observations made in our first pilot clinical trial (IND 8971, Study #1) that provided preliminary information on the safety and efficacy of immunotherapy with the anti-CD3 monoclonal antibody hOKT3γ1 (Ala-Ala), (currently called MGA031) combined with sirolimus and tacrolimus in preventing rejection and autoimmune destruction of deceased donor pancreatic islet transplants in type 1 diabetic recipients.

In the pilot study 4 of 6 single islet transplant recipients remained insulin independent with normal HbA1c and no episodes of hypoglycemia throughout the 1 year post-transplant period. Three of those four participants have maintained insulin independence for > 3.5, >4.5 and >5 years post islet transplant. These preliminary findings warrant an extension study involving more recipients and more comprehensive immunologic monitoring to examine in greater detail the impact of MGA031 induction immunotherapy on T cell responses operative in rejection and autoimmune destruction of transplanted islets as well as on formation of regulatory T cell function for the protection of transplanted islets.

A total of 5 patients with type 1 diabetes will be transplanted under this protocol. Islet transplant recipients will be admitted for 5 days and followed for one year after transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years of age.
2. Ability to provide written informed consent.
3. Mentally stable and able to comply with the procedures of the study.
4. Clinical history compatible with type 1 diabetes with onset of disease at <40 years of age and insulin-dependence for > 5 years at the time of enrollment.
5. Absent stimulated C-peptide (<0.3ng/ml) in response to a mixed meal tolerance test.
6. Involvement in intensive diabetes management defined as self monitoring of glucose values no less than a mean of three times each day averaged over each week and by the administration of three or more insulin injections each day or insulin pump therapy. Such management must be under the direction of an endocrinologist, diabetologist, or diabetes specialist with at least 3 clinical evaluations during the previous 12 months.
7. At least one episode of severe hypoglycemia in the past 3 years defined as an event with symptoms compatible with hypoglycemia in which the subject required the assistance of another person and which was associated with either a blood glucose level < 50 mg/dl or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration).
8. Reduced awareness of hypoglycemia.

Exclusion Criteria:

1. Any previous transplant.
2. BMI >27 kg/m2 or patient weight ≤ 50kg.
3. Insulin requirement of > 0.8 IU/kg/day or 50 IU/day.
4. HbA1c >10%.
5. Untreated proliferative diabetic retinopathy.
6. Uncontrolled Hypertension.
7. Estimated glomerular filtration rate <70 ml/min/1.73 m2 for females and <80 ml/min/1.73 m2 for males
8. Presence or history of macroalbuminuria (>300mg/d).
9. Presence or history of panel-reactive anti-HLA antibodies >20% by flow cytometry.
10. Females: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 3 months after discontinuation. Males: intent to procreate during the duration of the study or within 3 months after discontinuation or unwillingness to use effective measures of contraception.
11. Active infection.
12. Negative screen for Epstein-Barr Virus (EBV).
13. Invasive aspergillus infection within one year prior to study entry.
14. Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin.
15. Active alcohol, tobacco or substance abuse.
16. Baseline Hgb below the lower limits of normal at the local laboratory; lymphopenia, neutropenia, or thrombocytopenia.
17. A history of Factor V deficiency.
18. Any coagulopathy or medical condition requiring long-term anticoagulant therapy.
19. Severe co-existing cardiac disease.
20. Persistent elevation of liver function tests.
21. Symptomatic cholecystolithiasis.
22. Acute or chronic pancreatitis.
23. Symptomatic peptic ulcer disease.
24. Unremitting diarrhea, vomiting or other gastrointestinal disorders potentially interfering with absorption.
25. Hyperlipidemia despite medical therapy (fasting LDL cholesterol > 130 mg/dl, treated or untreated; and/or fasting triglycerides > 200 mg/dl).
26. Chronic use of systemic steroids.
27. Use of any other investigational agents within 4 weeks of participation.
28. Administration of live attenuated vaccine(s) within 2 months of enrollment.
29. Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-11; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard J. Hering, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Islet infusion with MGA031 induction and sirolimus and tacrolimus maintenance immunosuppression.
Period: Overall Study
Arm/Group | Experimental
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Full Islet Function.
Description: Proportion of subjects with full islet function (i.e. insulin independent) at one year after initial islet transplant.
Time Frame: At one year after initial transplant.
Population: The number of participants was based on the participants that were actually transplanted.
Measure: Number; unit: Participants
Groups:
- Experimental: Islet infusion
Arm/Group | Experimental
Number analyzed (Participants) | 5
Participants | 3

2. Primary Outcome: Serious Adverse Events Related to Immunosuppressive Therapy.
Description: Number of serious adverse events related to immunosuppressive therapy.
Time Frame: Day 0 - Day 365
Measure: Number; unit: Serious Adverse Events
Arm/Group | Experimental
Number analyzed (Participants) | 5
Serious Adverse Events | 0

3. Secondary Outcome: Subjects With Partial Islet Function and no Episodes of Severe Hypoglycemia;
Description: Proportion of subjects with partial islet function and no episodes of severe hypoglycemia at one year after initial islet transplant.
Time Frame: At one year after initial transplant
Measure: Number; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 5
Participants | 0

4. Secondary Outcome: Insulin Independent Single-donor Subjects.
Description: Proportion of insulin independent single-donor subjects at day 75 after transplant
Time Frame: At 75 days after transplant
Measure: Number; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 5
Participants | 1

5. Secondary Outcome: Insulin Independent Multiple-donor Subjects.
Description: Proportion of insulin independent multiple-donor subjects at one year after final transplant. Participant received more than one islet transplant.
Time Frame: At one year after final transplant
Measure: Number; unit: participants
Arm/Group | Experimental
Number analyzed (Participants) | 5
participants | 1

ADVERSE EVENTS:
Arm/Group | Experimental
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes